CLINICAL TRIAL: NCT01512043
Title: Breathing Control in Patients With Chronic Obstructive Pulmonary Disease (COPD) Intervention With Device-guided Breathing Control in COPD
Brief Title: Breathing Control in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lovisenberg Diakonale Hospital (Other)
Collaborators: University of Oslo (Other); Norwegian Foundation for Health and Rehabilitation (Other); University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2009/2/0285
Record Dates: First submitted 2011-12-08; First posted 2012-01-19 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: COPD
Keywords: Breathlessness; Symptoms; Quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1. Breathing control (Experimental): Description ...
  Interventions: Behavioral: Breathing control
- 2. Listening to music (Active Comparator): Listening to music without guiding on breathing on the same device as breathing control twice a day for four weeks. Using the device to measure breathing movements.
  Interventions: Behavioral: Breathing control
- 3. Silence (Sham Comparator): Using the device to measure breathing movement twice a day for four weeks. No instruction on breathing control and no music.
  Interventions: Behavioral: Breathing control

INTERVENTIONS:
Behavioral: Breathing control — Practice of device guided breathing control twice a day for four weeks.

SUMMARY:
There is a demand for explorative and comparative studies on various non-pharmaceutical efforts in treating and helping chronic obstructive pulmonary disease patients. This study has been developed in light of this need. The main purpose of the project is to test whether a device guided breathing control system can decreasing the feeling of breathlessness in patients with moderate stage and severe stage of COPD. In addition the study could shed light on whether a reduced feeling of breathlessness can lead to improved physical function, and less experience of other symptoms (I.e., depression, anxiety, sleeping difficulties, fatigue, pain) and provide a better quality of life for patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Dyspnoea symptoms in daily life
* Spirometry values showing a COPD moderate stage II (FEV1/FVC<70%, FEV1<80%) and severity grade at a severe stage III (FEV1/FVC<70%, FEV1<50% and FEV1 = 30% of a predicted)
* Be able to read, write and speak Norwegian
* Be at a stable phase of the disease

Exclusion Criteria:

* Changes in pulmonary medication during the last 4 weeks
* Diagnosis of cancer
* Presently attending a pulmonary rehabilitation course or other similar COPD education courses (due to the fact that these courses often have instructions on breathing control), or having attended similar courses during the last six months
* Ongoing exacerbation
* Attending other competitive studies
* Diagnosis of neuromuscular disease
* Diagnosis of dementia
* Attending help from a pulmonary physiotherapist

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Breathlessness | 4 months
  Questionnaires

SECONDARY OUTCOMES:
Depression | 4 months
  Questionnaires
Pulmonary functional tests | 4 months
Anxiety | 4 months
  Questionnaires
Fatigue | 4 months
  Questionnaire
Sleeping difficulties | 4 months
  Questionnaires
Pain | 4 months
  Questionnaire
6. Min walk test | 4 months
Arterial blood gas measures | 4 months
Quality of life | 4 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Astrid K Wahl, Professor, Principal Investigator — University of Oslo
Locations (1):
- Lovisenberg Diakonale Hospital, Oslo, Norway